CLINICAL TRIAL: NCT00602628
Title: WILL MULTIFUNCTIONAL MAGNETIC RESONANCE TECHNIQUES, DETAILED HISTOPATHOLOGICAL ANALYSIS AND PRONE TREATMENT POSITION IMPROVE ACCURACY OF TARGET VOLUME LOCALISATION & DEFINITION AND REDUCE EXPOSURE OF NORMAL TISSUES IN BREAST RADIOTHERAPY?
Brief Title: Radiation Therapy Planning Techniques in Reducing Damage to Normal Tissue in Women Undergoing Breast-Conserving Surgery for Ductal Carcinoma of the Breast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Diagnostic
Other Study IDs: RMH-CCR2981; CDR0000581130 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2008-01-24; First posted 2008-01-28 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2009-01

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ; invasive ductal breast carcinoma; breast cancer in situ; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Carcinoma, Ductal, Breast; Breast Carcinoma In Situ | interventions — Chemotherapy, Adjuvant; Biopsy; Magnetic Resonance Spectroscopy; High-Energy Shock Waves; Radiotherapy

INTERVENTIONS:
Other: questionnaire administration
Procedure: adjuvant therapy
Procedure: biopsy
Procedure: computed tomography
Procedure: dynamic contrast-enhanced magnetic resonance imaging
Procedure: magnetic resonance imaging
Procedure: therapeutic conventional surgery
Procedure: ultrasound imaging
Radiation: radiation therapy

SUMMARY:
RATIONALE: Diagnostic procedures, such as multifunctional magnetic resonance imaging and CT scans, may help reduce normal tissue damage in patients undergoing radiation therapy for cancer.

PURPOSE: This clinical trial is studying how well radiation therapy planning techniques work in reducing damage to normal tissue in women undergoing breast-conserving surgery for ductal breast carcinoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To improve precision of tumor bed localization and definition of clinical target volume, and to reduce normal tissue irradiation in women undergoing partial breast or breast boost radiotherapy.
* To test whether post-operative MRI improves the precision of tumor bed delineation after wide-local excision in comparison with the current standard CT scan/clip method.
* To determine the impact of tumor position within the excision specimen upon the localization of clinical target volume in relation to the tumor bed.
* To compare theoretical non-target tissue exposure from partial breast irradiation planned in the supine and prone (face-down) positions.

OUTLINE: Patients undergo planned breast-conservation surgery and placement of titanium clips to the four radial, the deep, and superficial margins of the excision cavity (for localization of tumor bed).

Within 2 weeks after surgery, patients undergo supine radiotherapy-planning CT scan as standard analysis. Patients then undergo a radiotherapy-planning CT scan in the prone position. Patients complete a linear analogue questionnaire after both scans designed to assess patient comfort and anxiety in each position. Patients then undergo multifunctional MRI (including dynamic contrast-enhancement MRI and diffusion-weighted MRI) of the ipsilateral breast in the prone position (≥ 3 weeks after surgery). If suspicious lesions ≥ 5 mm are found on MRI, patients are referred for a second-look ultrasound with biopsy (if lesion visible on ultrasound); where suspicious lesions are seen only on MRI, patients undergo MRI-guided biopsy. Lesions < 5 mm are included in the whole-breast radiotherapy treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Planning to undergo breast-conserving surgery (BCS)* for unifocal ductal carcinoma in situ (DCIS) or grade 1-2 invasive ductal carcinoma (IDC) of the breast NOTE: *Patients who have underwent BCS and have titanium clips placed according to this protocol are eligible for this study.
* No T4d or multifocal disease (as defined on mammography or ultrasound)
* No G3 disease
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Female
* Menopausal status not specified

Exclusion criteria:

* Cup size DD or greater
* Ferromagnetic implants (exclude participation in MRI)
* Claustrophobia (exclude participation in MRI)
* Gadolinium allergy

PRIOR CONCURRENT THERAPY:

* No prior surgery to ipsilateral breast
* No prior neoadjuvant chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-07 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Difference in lung NTDmean (biologically weighted [normalized] mean of total dose to lung normalized to 2 Gy fractions) in supine vs prone positions

SECONDARY OUTCOMES:
Closeness of agreement between MRI-based vs CT scan/clip- based delineation of tumor bed
Closeness of agreement between clinical target volumes (CTVs) defined using uniform margin vs those defined using knowledge of all excision margins
Difference in NTDmean to ipsilateral non-planning target volume (PTV) breast tissue, chest wall muscle, and heart
Difference in mean volume of PTV in supine versus prone positions
Difference in dose homogeneity within PTV in each position
Difference in complexity of beams needed to achieve above dose homogeneity within PTV
Patient comfort with each positioning technique (assessed by questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: John R. Yarnold, MD, FRCR, Study Chair — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden - Surrey, Sutton, England, United Kingdom